CLINICAL TRIAL: NCT05139082
Title: A Phase I/II Phase Evaluating the Effectiveness and Safety of CDK4/6 Inhibitor (TQB3616) Combined With PD-L1 Monoclonal Antibody (TQB2450) in the Treatment of PD-1/PD-L1 Monoclonal Antibody Resistance and Abnormal Cell Cycle Digestive System Tumors.
Brief Title: Study of CDK4/6 Inhibitor Combined With PD-L1 Monoclonal Antibody in the Treatment of PD-1/PD-L1 Resistance and Abnormal Cell Cycle Digestive System Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Beijing Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3616-TQB2450-I/II-01
Record Dates: First submitted 2021-11-11; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Digestive System Tumors
Keywords: PD-1/PD-L1 resistance; abnormal cell cycle

STUDY DESIGN:
Intervention Model Description: PD-1/PD-L1 monoclonal antibody resistance, abnormal cell cycle, digestive system tumors
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDK4/6 inhibitor (TQB3616) + PD-L1 monoclonal antibody (TQB2450) (Other): TQB3616 capsules (120/150/180mg p.o. qd, d1-d21) combined with TQB2450 injection (1200mg ivgtt, d1)
  Interventions: Drug: TQB3616 capsules＋ TQB2450 injection

INTERVENTIONS:
Drug: TQB3616 capsules＋ TQB2450 injection — TQB3616 is a highly active CDK4/6 inhibitor. Preclinical studies have shown that it has a strong inhibitory effect on the kinase activity of CDK4/6.
  TQB2450 is a humanized monoclonal antibody targeting PD-L1, which prevents PD-L1 from binding to the PD-1 and B7.1 receptors on the surface of T cells, so as to restore the activity of T cells and thereby enhance the immune response, and has the potential to treat various types of tumors.

SUMMARY:
This study intends to explore the effectiveness and safety of CDK4/6 inhibitor (TQB3616) combined with PD-L1 monoclonal antibody (TQB2450) in the treatment of PD-1/PD-L1 monoclonal antibody resistance and abnormal cell cycle digestive system tumors, through prospective Explore to provide more evidence-based medical evidence for precision immunotherapy for patients with digestive system tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent;
2. Age ≥ 18 years old;
3. No gender limitation;
4. Digestive system malignant tumor diagnosed by pathology;
5. Digestive system tumor patients who have failed standard treatment;
6. Patients with PD-1 monoclonal antibody or PD-L1 monoclonal antibody treatment failure;
7. Abnormal cell cycle signaling pathways
8. Patients with unresectable digestive system tumors confirmed by imaging;
9. There is at least one measurable lesion (according to the RECIST1.1 standard) or an unmeasurable lesion that can be evaluated, and the imaging diagnosis is ≤21 days from the selection time；
10. The expected survival period is ≥3 months;
11. General physical status (ECOG) 0-2;
12. Sufficient bone marrow hematopoietic function (within 7 days);
13. Heart, lung, kidney, and liver functions are generally normal.
14. Women of childbearing age should agree to use effective contraceptive measures during the study period and 6 months after the end of the study, and have a negative serum or urine pregnancy test within 7 days before enrollment in the study; men should agree to use effective contraception during the study period and after the end of the study period 6 Effective contraceptive measures must be used within one month.

Exclusion Criteria:

1. People who are currently receiving other effective treatments;
2. Patients who are using immunosuppressive agents or systemic or absorptive local hormone therapy to achieve immunosuppression within 2 weeks before the first medication;
3. Patients who have participated in other clinical trials within 4 weeks before enrollment;
4. Allergic to study drugs; 5 . Those without measurable tumor lesions, such as body cavity effusion or diffuse infiltration of organs;

6. Those with measurable lesions that have received radiotherapy. 7. Patients with other primary malignant tumors other than digestive system tumors at the same time, except for early solid tumors that have been cured for more than 1 year; 8. Clinically significant cardiovascular diseases, such as heart failure (NYHAIII-IV), are not controlled A history of coronary heart disease, cardiomyopathy, arrhythmia, uncontrolled hypertension or myocardial infarction within the past 1 year; 9. Neurological or mental disorders that affect cognitive ability, including central nervous system metastasis; 10. Existed within 14 days before enrollment Active severe clinical infections (>grade 2 NCI-CTCAE version 5.0), including active tuberculosis; 11. Known or self-reported HIV infection or active hepatitis B or C; 12. Uncontrolled Systemic diseases, such as poorly controlled diabetes; 13. A history of interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or evidence of interstitial lung disease on baseline chest X-ray/CT; 14. Keratitis , Ulcerative keratitis or severe dry eye; 15. Known hypersensitivity or allergic reaction to any component of the study drug; 16. Pregnancy (determined by serum β-chorionic gonadotropin test) or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-24 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 48 weeks
  Objective response rate refers to the percentage of complete (CR) or partial response (PR) subjects determined by the investigator based on RECIST 1.1 or iRECIST (CR under iRECIST criteria, PR can occur after imaging disease progression).

SECONDARY OUTCOMES:
Disease control rate（DCR） | up to 48 weeks
  Disease control rate refers to the percentage of subjects with complete remission, partial remission, or stable disease (SD) of 6 weeks or more as determined by RECIST 1.1 or iRECIST (CR, PR, SD under iRECIST criteria can occur after imaging disease progression).
Overall survival (OS) | up to 48 weeks
  Overall survival defined as the time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: lin shen, master, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No